CLINICAL TRIAL: NCT03610919
Title: Effects of Oxytocin Dose Frequency on Behavioral and Neural Responses, and Modulation by Trait Autism and Genotype
Brief Title: Effects of Oxytocin Dose Frequency on Behavioral and Neural Responses
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-57
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: multiple doses; oxytocin; genotype; autism trait
MeSH Terms: interventions — Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin nasal spray(5 doses) (Experimental): Oxytocin nasal spray for 5 days, 24 IU per day
  Interventions: Drug: Nasal Sprays
- Oxytocin nasal spray(3 doses) (Experimental): Oxytocin nasal spray or placebo nasal spray interleaved during the 5 days( on the 1st,3rd and 5th day),24 IU per day.
  Interventions: Drug: Nasal Sprays
- Placebo nasal spray(control group) (Placebo Comparator): Placebo nasal spray for 5 days,24 IU per day.
  Interventions: Drug: Nasal Sprays

INTERVENTIONS:
Drug: Nasal Sprays — Intranasal administration of 24 international units per dose.

SUMMARY:
The main aim of the study is to examine effects of different dose frequencies of repeated oxytocin administration on neural and behavioral markers of oxytocin in healthy male subjects. In addition modulatory effects of autism traits and oxytocin receptor genotype (OXTR) will be explored.

DETAILED DESCRIPTION:
In the present study, healthy male subjects will be screened according to the study inclusion criteria. After enrollment buccal swaps will be collected for genotyping and subjects will be randomly assigned to three experimental groups that will receive treatment for 5 subsequent days: (1) placebo for five days, (2) oxytocin on days 1, 3 and 5, or (3) oxytocin for five days. Behavioral measures, task-based and resting fMRI will be assessed after the first treatment (acute effects) and the last treatment (chronic effects). The task-based fMRI will employ an implicit emotional face processing paradigm and ratings of the facial emotions will be collected after the fMRI.

Moreover, to control for potential confounding effects of relevant traits all participants will complete the following questionnaires: Interpersonal Reactivity Index (IRI),Beck depression inventory (BDI), State-Trait Anxiety Inventory (STAI). To explore potential modulatory effects of trait autism, all subjects will be administered the Autism Spectrum Quotient (ASQ) scale to assess pre-treatment autism traits.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult males

Exclusion Criteria:

* past or current psychiatric or neurological disorder head trauma substance abuse medication fMRI contraindications (e.g. metal implants)

Ages: 17 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Between group differences in the changes between acute and chronic administration effects of oxytocin on amygdala reactivity towards fearful faces as assessed by fMRI. | 45 minutes after treatment (day 1 vs day 5)
  Differences between the treatment groups will be determined by examining differential changes of acute treatment (day 1) vs chronic treatment (day 5) on amygdala activity towards fearful faces. Amygdala activity will be assessed using task-based BOLD fMRI analyses.
Between group differences in the changes between acute and chronic administration effects of oxytocin on amygdala resting state connectivity as assessed by fMRI. | 45 minutes after treatment (day 1 vs day 5)
  Differences between the treatment groups will be determined by examining differential changes of acute treatment (day 1) vs chronic treatment (day 5) on amygdala resting state fMRI connectivity. Amygdala functional connectivity will be examined using a seed to whole brain approach.

SECONDARY OUTCOMES:
Association between trait autism with acute and chronic treatment effects on amygdala activity in response to fearful faces | 45 minutes after treatment (day 1 vs day 5)
  Associations between autism traits and amygdala response to fearful faces during acute effects (single dose, day 1) and chronic effects (over the course of 5 days) will be examined by means of correlation analyses. Pre-treatment autism trait scores will be assessed using the Autism Spectrum Quotient (ASQ)
Association between trait autism with acute and chronic treatment effects on amygdala resting state connectivity | 45 minutes after treatment (day 1 vs day 5)
  Associations between autism traits and amygdala resting state connectivity during acute effects (single dose, day 1) and chronic effects (over the course of 5 days) will be examined by means of correlation analyses. Pre-treatment autism trait scores will be assessed using the Autism Spectrum Quotient (ASQ)
Interaction of acute and chronic treatment effects on amygdala activity with oxytocin receptor genotype. | 45 minutes after treatment (day 1 vs day 5)
  Participants will be divided in sub-groups according to their oxytocin receptor (OXTR) genetic profile. Modulatory effects of the OXTR on acute and chronic effects will be explored by comparing effects of treatment on amygdala activity in response to fearful faces as assessed by fMRI between the genotype groups.
Interaction of acute and chronic treatment effects on amygdala connectivity with oxytocin receptor genotype. | 45 minutes after treatment (day 1 vs day 5)
  Participants will be divided in sub-groups according to their oxytocin receptor (OXTR) genetic profile. Modulatory effects of the OXTR on acute and chronic effects will be explored by comparing effects of treatment on amygdala resting state connectivity as assessed by fMRI between the genotype groups.
Treatment effects on arousal will be assessed by subjects rating their arousal on a 9-point Likert scale in response to the face pictures presented again after their fMRI scans on day 1 and day 5 | 45 minutes after treatment (day 1 vs day 5)
  After assessment of the implicit fMRI emotional face paradigm participants will rate the emotional arousal of the stimuli using Likert scales (9 point). Acute and chronic effects will be assessed using repeated measures ANOVAs (day 1 vs day 5) to compare differential changes between the groups.
Treatment effects on valence will be assessed by subjects rating their valence on a 9 point Likert scale in response to the face pictures presented again after their fMRI scans on day 1 and day 5 | 45 minutes after treatment (day 1 vs day 5)
  After assessment of the implicit fMRI emotional face paradigm participants will rate the emotional valence of the stimuli using Likert scales (9 point). Acute and chronic effects will be assessed using repeated measures ANOVAs (day 1 vs day 5) to compare differential changes between the groups.
Treatment effects on intensity will be assessed by subjects rating their intensity on a 9 point Likert scale in response to the face pictures presented again after their fMRI scans on day 1 and day 5 | 45 minutes after treatment (day 1 vs day 5)
  After assessment of the implicit fMRI emotional face paradigm participants will rate the emotional intensity of the stimuli using Likert scales (9 point). Acute and chronic effects will be assessed using repeated measures ANOVAs (day 1 vs day 5) to compare differential changes between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- school of life science and technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China